CLINICAL TRIAL: NCT02950818
Title: A Partnership to Translate an Evidence-based Intervention for Vulnerable Older Adults With Heart Disease
Brief Title: A Partnership to Translate an Evidence-based Intervention (Take Heart) for Vulnerable Older Adults With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Detroit Medical Center (Other); Detroit Area Agency on Aging (Other)
Responsible Party: Principal Investigator, Cathleen M Connell, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00092196; 1R01AG047203-01A1 (NIH)
Record Dates: First submitted 2016-04-01; First posted 2016-11-01 (Estimated); Results first posted 2022-08-25 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: Heart Diseases
Keywords: self-care; health education; chronic disease; heart diseases; risk factors for heart disease
MeSH Terms: conditions — Heart Diseases; Health Education; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take Heart self-management program (Experimental): Group and telephone-based educational program to enhance self-management of heart disease and related risk factors.
  Interventions: Behavioral: Take Heart
- Waitlist control (No Intervention): Control group participants will be offered the opportunity to participate in Take Heart following the conclusion of their study involvement.

INTERVENTIONS:
Behavioral: Take Heart — Participants receive an evidence-based heart disease self management program consisting of a combination of five two and a half hour group sessions and telephone counseling offered by a trained facilitator employed by the Detroit Area Agency on Aging. The program is designed so that participants select an area to work on (e.g., diet, exercise, medication taking, communication with health care professionals) and receive support, information, and encouragement from group members and program facilitators, to help them reach their goals.
  Arms: Take Heart self-management program

SUMMARY:
To evaluate the effectiveness of Take Heart, a behavioral/educational program for adults age 50+ with heart disease, or with at least two risk factors for heart disease, that helps them to better manage their health condition(s). Take Heart is a new version of an evidence-based program that has recently been adapted to be suitable for the needs of adults residing in Detroit.

DETAILED DESCRIPTION:
In this study, a heart disease self-management program will be tested in a low-income, predominantly African-American community via a partnership with the Detroit Area Agency on Aging (DAAA), the Detroit Medical Center (DMC), and University of Michigan School of Public Health's Center for Managing Chronic Disease (CMCD). The specific aims of the research are to: (1) adapt existing program materials to be appropriate for the new target population, getting feedback from various sources including focus group interviews; (2) conduct a pilot study of the adapted "Take Heart" program; (3) refine the intervention and conduct a randomized trial with 376 participants age 50 years and over, to assess health outcomes; (4) assess the translation and implementation of the intervention in the target setting and identify factors that help and hinder the process; (5) assess cost savings associated with the intervention; and (6) develop guidelines for "scaling up", that is, for replicating the program in other low-income areas through the national network of Area Agencies on Aging.

ELIGIBILITY:
Inclusion criteria:

50 years or older

1 or more diagnosed cardiovascular conditions, including:

* Atrial fibrillation
* Angina
* Myocardial infarction
* Congestive heart failure
* Valvular disease (aortic stenosis or mitral regurgitation)
* Peripheral vascular disease
* Pulmonary hypertension
* OR >2 major risk factors for cardiovascular disease (CVD; high cholesterol, high blood pressure, smoking, diabetes, chronic kidney disease-stage 3 or 4)
* Must have access to a mobile or landline telephone
* Must be able to travel to group sessions, with or without transportation assistance

Exclusion Criteria

• Limited fluency in English posing significant barrier to deriving program benefit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen M Connell, PhD, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan, School of Public Health, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing: We will have self-reported data (baseline and 12-month) on health, demographics, and psychosocial functioning from both intervention and control participants. An anonymized dataset will be created, which will be made available to other researchers who have appropriate approvals from all relevant Institutional Review Boards (IRBs) through a secure file transfer protocol (FTP) site, M+Box, whose encryption protocols allow secure uploading of files, with sharing limited to specified users (see: http://www.itcs.umich.edu/storage/box/faq.php#storage). Data dictionaries and data collection forms will also be made available. Researchers using the data will be instructed to delete their copy of the dataset once analyses are complete. An email address to reach University of Michigan investigators will be available for questions about the datasets.

REFERENCES:
- [Derived] Janevic MR, Ramsay JE, Allgood KL, Domazet A, Cardozo S, Connell CM. Heart Disease Self-management for African American Older Adults: Outcomes of an Adapted Evidence-Based Intervention. Innov Aging. 2022 Aug 19;6(7):igac053. doi: 10.1093/geroni/igac053. eCollection 2022. PMID 36267321

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Take Heart Self-management Program | Waitlist Control
Started | 228 | 225
Completed | 161 | 201
Not Completed | 67 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Take Heart Self-management Program | Waitlist Control | Total
Number analyzed (Participants) | 228 | 225 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (9.3) | 65.3 (8.6) | 65.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We had missing data on sex for one participant.
  Participants
    number analyzed (Participants) | 228 | 224 | 452
    Female | 155 | 179 | 334
    Male | 73 | 45 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 203 | 197 | 400
  Unknown or Not Reported | 23 | 26 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 193 | 187 | 380
  White | 10 | 10 | 20
  More than one race | 20 | 21 | 41
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 228 | 225 | 453
Education [Count of Participants; unit: Participants] — Population: Missing education data on participants.
  Participants
    number analyzed (Participants) | 226 | 225 | 451
    <High School | 23 | 30 | 53
    High School Grad or GED | 55 | 56 | 111
    Some College | 107 | 87 | 194
    College Graduate or Higher | 41 | 52 | 93
Marital Status [Count of Participants; unit: Participants] — Population: Missing data on participants.
  Participants
    number analyzed (Participants) | 224 | 225 | 449
    Married/Partnered | 24 | 33 | 57
    Single | 200 | 192 | 392
Employment Status [Count of Participants; unit: Participants] — Population: Missing data on some participants.
  Participants
    number analyzed (Participants) | 224 | 225 | 449
    Employed | 26 | 19 | 45
    Retired | 107 | 119 | 226
    Unemployed | 45 | 41 | 86
    Other | 46 | 46 | 92
Self-Rated Health [Count of Participants; unit: Participants] — Population: Missing data on participant.
  Participants
    number analyzed (Participants) | 227 | 225 | 452
    Excellent | 2 | 6 | 8
    Very Good | 22 | 19 | 41
    Good | 79 | 67 | 146
    Fair | 89 | 88 | 177
    Poor | 35 | 45 | 80
Heart Disease Diagnoses [Number; unit: participants]
  Atrial Fibrilation | 42 | 44 | 86
  Myocardial Infarction | 41 | 38 | 79
  Valvular Disease | 12 | 22 | 34
  Pulmonary Hypertension | 11 | 7 | 18
  Angina | 33 | 44 | 77
  Congestive Heart Failure | 33 | 45 | 78
  Peripheral Vascular Disease | 27 | 26 | 53
  Other Heart Disease Condition | 9 | 6 | 15
Heart Disease Risk Factors [Number; unit: participants]
  High Cholesterol | 184 | 170 | 354
  High Blood Pressure | 210 | 204 | 414
  Diabetes | 109 | 88 | 197
  Chronic Kidney Disease | 10 | 16 | 26
  Current Smoker | 63 | 70 | 133
Comorbidities [Number; unit: particiapnts]
  Depression | 91 | 80 | 171
  Cancer | 35 | 35 | 70
  Prediabetes | 104 | 84 | 188
  Stroke | 33 | 42 | 75
  Arthritis | 146 | 158 | 304
  COPD | 50 | 71 | 121
  Asthma | 57 | 64 | 121
Healthcare Utilization - ED Visits [Mean (Standard Deviation); unit: ED Visits in past 12 months] | 1.3 (1.7) | 1.7 (3.9) | 1.5 (3.1)
PROMIS-29 [Mean (Standard Deviation); unit: units on a scale] — PROMIS-29 measures 8 domains of health-related qualify of life among adults.Domains have 4 items ranked on Likert scales: physical functioning, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles/activities, pain interference, pain intensity.All domains except pain intensity, raw subscale are summed and converted to T-scores (standardized score, mean 50, SD 10) using HealthMeasures.net conversion tables, lower=better.Pain intensity measured on11 point scale (0 -10, 0=no pain, 10=worst pain).T-score rescales raw score into standardized score, mean 50, SD 10.
  units on a scale
    Physical Functioning | 33.1 (6.8) | 34.5 (7.1) | 33.9 (7)
    Anxiety | 53.7 (9.4) | 54.1 (9.7) | 53.9 (9.5)
    Depression | 50.3 (8.2) | 51.2 (9.3) | 50.8 (8.8)
    Fatigue | 51.8 (9.3) | 53.5 (9.7) | 52.7 (9.5)
    Sleep | 51.9 (3.3) | 52.4 (3.6) | 52.2 (3.5)
    Social | 38.9 (9.1) | 38.8 (8.6) | 38.8 (8.8)
    Pain Interference | 57.3 (10.1) | 58.8 (10) | 58.1 (10.1)
    Pain Intensity | 4.9 (2.6) | 5.5 (2.7) | 5.3 (2.7)
Heart Related Symptoms [Mean (Standard Deviation); unit: symptoms] — The cardiac symptom subscale of the Symptom and Health Problem Profile (Janz et al.,1999) asks about the frequency of chest pain/discomfort; shortness of breath; waking up from sleep because of chest pain or pressure; waking up from sleep because of shortness of breath or difficulty breathing; and irregular heartbeat or palpitations (not present, once or twice/week, a few times/week, once/day, several times/day) in the prior 12 months. Symptom frequency (0 to 4) was summed, yielding an overall symptom burden score that ranged from 0 to 20 (higher is worse). Means are reported.
  symptoms | 1.3 (1.5) | 1.7 (1.5) | 1.5 (1.5)
Healthcare Utilization - Hospitalizations [Mean (Standard Deviation); unit: Hospitalizations in past 12 months] | 1.8 (5) | 2.4 (9.3) | 2.1 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Hospitalizations
Description: This will be measured by asking participants to report the number of nights they have stayed overnight in the hospital during the past year, for something related to their own health. We will ask this at baseline and then at the 12 month mark after the completion of the baseline survey, so that we can compare the year prior to the intervention to the year they completed the intervention. In addition, when possible, we will verify self-reported hospitalizations with Electronic Medical Record (EMR) data from our partners at the Detroit Medical Center (DMC). We will only be able to look into the EMRs of those participants that are patients at the DMC. Change will be indicated by difference between count at baseline and count at follow-up.
Time Frame: Baseline and 12-month follow up
Measure: Mean (95% Confidence Interval); unit: hospitalizations
Arm/Group | Take Heart Self-management Program | Waitlist Control
Number analyzed (Participants) | 161 | 201
hospitalizations | 0.98 [0.98 to 1.6] | 1.48 [1.19 to 1.84]

2. Primary Outcome: Emergency Department Visits
Description: This will be measured by asking participants to report the number of times they went to the emergency department for something related to their own health, during the past year. We will ask this at baseline and then at the 12 month mark after the completion of the baseline survey, so that we can compare the year prior to the intervention to the year they completed the intervention. In addition, when possible, we will verify self-reported Emergency Department visits with Electronic Medical Record (EMR) data from our partners at the Detroit Medical Center (DMC). We will only be able to look into the EMRs of those participants that are patients at the DMC. Change will be indicated by difference between count at baseline and count at follow-up.
Time Frame: Baseline and 12 month follow up
Measure: Mean (95% Confidence Interval); unit: ED visits
Arm/Group | Take Heart Self-management Program | Waitlist Control
Number analyzed (Participants) | 161 | 201
ED visits | 2.55 [1.64 to 3.97] | 2.74 [1.76 to 4.27]

3. Secondary Outcome: Health-related Quality of Life
Description: Health-related quality of life (HRQOL) was measured with the PROMIS-29 (Patient-Reported Outcomes Measurement Information System-29) profile measure, which assesses depression, anxiety, pain interference, physical function, fatigue, satisfaction with social role participation, and sleep disturbance (4 items each, 5 point Likert scales). Higher values indicate poorer health. One item (11 point scale) measures pain intensity on a scale of 0 -10, 0=no pain, 10=worst pain). The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. https://www.assessmentcenter.net/documents/PROMIS%20Profile%20Scoring%20Manual.pdf This table indicates the mean score in each domain at the 12-month follow up time point for both intervention and control groups, as well as the difference between the means of the two groups at the 12-month time point.
Time Frame: Baseline and 12-month follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Means Difference Between Groups: Means differences at 12 months between intervention and control groups (Intervention minus control)
Arm/Group | Take Heart Self-management Program | Waitlist Control | Means Difference Between Groups
Number analyzed (Participants) | 161 | 201 | 362
units on a scale
  Physical Functioning | 33 [31.9 to 34.2] | 34.1 [33 to 35.2] | -1.1 [-2.446 to 0.297]
  Anxiety | 54.1 [52.5 to 55.7] | 54.1 [52.6 to 55.6] | 0.001 [-1.907 to 1.910]
  Depression | 51 [49.4 to 52.6] | 51.3 [49.8 to 52.7] | -0.26 [-2.116 to 1.600]
  Fatigue | 51.3 [49.8 to 52.9] | 54.2 [52.7 to 55.6] | -2.82 [-4.697 to -0.947]
  Sleep | 51.9 [51.3 to 52.5] | 52.6 [52.1 to 53.2] | -0.727 [-1.431 to -0.023]
  Social | 38.9 [34.4 to 40.5] | 40.1 [28.6 to 41.5] | -1.129 [-2.977 to 0.718]
  Pain Interference | 57.6 [55.8 to 59.4] | 58.9 [57.2 to 60.6] | -1.332 [-3.467 to 0.802]
  Pain Intensity | 5.1 [4.6 to 5.5] | 5.4 [4.9 to 5.8] | -0.318 [-0.854 to 0.218]

4. Secondary Outcome: Cardiac Symptom Experience
Description: The cardiac symptom subscale of the Symptom and Health Problem Profile (Janz et al., 1999) asks about the frequency of chest pain/discomfort; shortness of breath; waking up from sleep because of chest pain or pressure; waking up from sleep because of shortness of breath or difficulty breathing; and irregular heartbeat or palpitations (not present, once or twice/week, a few times/week, once/day, several times/day) in the prior 12 months. Symptom frequency (0 to 4) was summed, yielding an overall symptom burden score that ranged from 0 to 20. Higher scores indicate worse health. Change is indicated by the difference in mean frequency from baseline to follow-up.
Time Frame: Baseline and 12-month follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Take Heart Self-management Program | Waitlist Control
Number analyzed (Participants) | 161 | 201
units on a scale | 1.96 [1.35 to 2.58] | 2.74 [2.17 to 3.32]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from baseline through study completion, an average of 1 year.
Arm/Group | Take Heart Self-management Program | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 1/228 | 1/225
Serious Adverse Events (participants affected / at risk) | 7/228 | 0/225
Other Adverse Events (participants affected / at risk) | 0/228 | 0/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Take Heart Self-management Program (N=228) | Waitlist Control (N=225)
ED Visit (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Heart Attack (Cardiac disorders) | 4 | 0
Stroke (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02950818/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT02950818/ICF_001.pdf